CLINICAL TRIAL: NCT00877045
Title: Treatment Patterns in Gastrointestinal Stromal Tumors in the Community Oncology Setting
Status: Completed | Type: Observational
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Jeffrey F. Patton, M.D., SCRI Oncology Research Consortium
Other Study IDs: SCRI OUTCOMES 01
Record Dates: First submitted 2009-04-03; First posted 2009-04-07 (Estimated); Last update posted 2010-08-04 (Estimated); Status verified 2010-08

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: Gastrointestinal Stromal Tumors; GIST; tyrosine kinase inhibitors; Imatinib; Gleevec; Suntinib; Sutent
MeSH Terms: conditions — Gastrointestinal Stromal Tumors

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
This is a retrospective medical record abstraction to evaluate the patterns of care for Gastrointestinal stromal tumors (GIST) in the community setting. Patient demographics and characteristics along with the treatments received will be described. Investigators will establish the percentage of patients who undergo surgery, the percentage of patients who are treated with kinase inhibitors as well as in what setting (adjuvant or metastatic) as well as the duration of therapy. Physician information will also be collected to assess for differences in treatment based on physician or geographical differences.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with GIST based on ICD-9 code from January 2005 to present will be eligible. This will include current active patients as well as patients who have expired and have medical chart available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients diagnosed with GIST based on ICD-9 code from January 2005 to present will be eligible. This will include current active patients as well as patients who have expired and have medical chart available. Estimate reviewing approximately 300 charts total.
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2008-01; Primary Completion 2009-01 (Actual); Study Completion 2009-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey F Patton, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (5):
- United States (5):
  - Florida Cancer Specialists, Fort Myers, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, PLLC, Nashville, Tennessee
  - Virginia Cancer Institute, Richmond, Virginia